CLINICAL TRIAL: NCT02787408
Title: The SPACER Trial - Repair of Tricuspid Valve Regurgitation Using the Edwards TricuSPid TrAnsCatheter REpaiR System
Acronym: SPACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-09
Record Dates: First submitted 2016-04-11; First posted 2016-06-01 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-04

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EW Tricuspid Transcatheter Repair System (Experimental): Edwards (EW) Tricuspid Transcatheter Repair System
  Interventions: Device: EW Tricuspid Transcatheter Repair System

INTERVENTIONS:
Device: EW Tricuspid Transcatheter Repair System — Treatment with the EW Tricuspid Transcatheter Repair System

SUMMARY:
The purpose of the study is to assess the safety and device performance of the Edwards Tricuspid Transcatheter Repair System in patients with clinically significant, symptomatic, tricuspid regurgitation who are at high surgical risk for standard tricuspid repair/replacement.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety and device performance of the Edwards Tricuspid Transcatheter Repair System in patients with clinically significant, symptomatic, tricuspid regurgitation who are at high surgical risk for standard tricuspid repair/replacement. The study is a multi-center, international, prospective, single arm, safety study. Enrolled subjects will be assessed for clinical follow-up at 1 month, 6 months, 1 year and annually for 3 years post implant procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Ethics Committee (EC) approved study consent form prior to study related procedures
2. Eighteen years of age or older
3. Clinically significant, symptomatic (New York Heart Association (NYHA) Functional Class II or greater), tricuspid regurgitation (per applicable guidelines) requiring tricuspid valve repair or replacement as assessed by the Heart Team
4. Functional tricuspid regurgitation as the primary etiology
5. New York Heart Association (NYHA) Functional Class II or greater or signs of persistent right heart failure despite optimal medical therapy
6. Determined by the 'HEART Team' (a minimum of one Cardiologist, and one Cardiac Surgeon) to be at high surgical risk for tricuspid valve repair or replacement and the benefit-risk analysis supports utilization of the investigational device
7. Willing to attend study follow-up assessments for up to 3 years

Exclusion Criteria

1. Tricuspid valve/right heart anatomy not suitable for the study device:

   1. Native tricuspid annulus area < 2.14 cm2 (9 mm device) or < 2.63 cm2 (12 mm device) or < 3.27cm2 (15 mm device) as measured by transthoracic echocardiography
   2. Sub-valvular structures/anatomy that would preclude from proper anchor or coaptation device placement, positioning and retrieval
   3. Access pathway vessel diameter less than 7.1 mm (9, 12 mm and 15 mm devices)
2. Moderate or greater tricuspid valve stenosis
3. Untreated clinically significant coronary artery disease requiring immediate revascularization
4. Any therapeutic invasive cardiac procedure performed within 30 days of the scheduled implant procedure
5. Patients not already receiving dialysis with renal insufficiency (eGFR <25) per lab test ≤ 48 hours prior to scheduled implant procedure
6. Myocardial infarction within 30 days of scheduled implant procedure
7. Hemodynamic instability within 30 days of scheduled implant procedure
8. Patient requiring surgery under general anesthesia for any reason within 90 days of scheduled implant procedure
9. Severe left ventricular dysfunction with ejection fraction < 25% within 90 days of scheduled implant procedure
10. Patients with pulmonary artery systolic pressure > 70 mmHg via transthoracic echocardiography or alternative standard modality (e.g., direct pressure measurement) within 90 days
11. Concomitant clinically significant valve (aortic, mitral, or pulmonic) disease requiring immediate (± 30 days of study procedure) repair or replacement
12. Active endocarditis or infection within 3 months of scheduled implant procedure
13. Cerebrovascular accident within 3 months of scheduled implant procedure
14. Non-cardiac disease limiting life expectancy to be less than 12 months at baseline evaluation
15. Documented history of bleeding diathesis, coagulopathy or gastrointestinal bleeding within 3 months of scheduled implant procedure
16. Evidence of right sided intracardiac mass, thrombus, or vegetation
17. Prior venous stent placed within the access route (e.g., sub-clavian vein) that could negatively react with device
18. Previously treated tricuspid valve which included implantation of a bioprosthetic valve or mechanical valve
19. Known hypersensitivity to cobalt chromium, nitinol or titanium
20. Known hypersensitivity to anticoagulation therapy or contrast agent, which cannot be adequately medicated
21. Patient is a current intravenous drug user
22. Female of child-bearing potential is pregnant or lactating
23. Patient is currently participating or has participated in another investigational drug or device clinical study within 30 days of study screening activity
24. Patient requires emergent/emergency treatment for tricuspid insufficiency
25. Patient is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (3):
  - St. Paul's Hospital, Providence Health Care Research Institute, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec-Universite Laval, Québec
- France (2):
  - Institut Hospitalier Jacques Cartier, Massy
  - Hōpital Charles Nicolle, Rouen
- Germany (4):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Charite-Universitätsmedzin Berlin, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - Munich University Clinic, Ludwig-Maximilian University, Munich
- Hygeia Hospital, Athens, Greece
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EW Tricuspid Transcatheter Repair System
Started | 25
Completed | 7
Not Completed | 18
Not completed — Death | 16
Not completed — Withdrawal by Subject | 1
Not completed — Non-implanted patient exited post 6 month follow-up visit per protocol | 1

BASELINE CHARACTERISTICS:
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 4
  Canada | 11
  France | 1
  Switzerland | 1
  Germany | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4.74)
New York Heart Association Class (NYHA) [Count of Participants; unit: Participants] — Measure Description: NYHA Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    Class I | 0
    Class II | 6
    Class III | 14
    Class IV | 5
The European System for Cardiac Operative Risk Evaluation: EuroScore II [Mean (Standard Deviation); unit: Percentage of surgical risk] — Measure Description:
  The European System for Cardiac Operative Risk Evaluation (EuroScore II) is a risk model which allows the calculation of the risk of death after a heart operation. The higher the score percentage, the higher the risk of an adverse outcome.
  The EuroScore II Scale ranges from 0-100%. Although the maximum value of the full range is 100%, any percentage over 10 is considered a high risk for surgical mortality.
  EuroScore II risk levels are as follows:
  < 8%: Low risk
  8-10%: Moderate risk
  >10%: High risk
  Percentage of surgical risk | 11.5 (7.65)
History of Heart Failure [Count of Participants; unit: Participants] | 13
Hospitalization for Heart Failure prior 6 months [Count of Participants; unit: Participants] | 13
Diabetes [Count of Participants; unit: Participants]
  No | 22
  Type 1 | 0
  Type II ( Insulin treated) | 1
  Type II ( Non-Insulin treated) | 2
Cancer [Count of Participants; unit: Participants] | 3
Carotid Artery Disease [Count of Participants; unit: Participants] | 2
Coagulopathy [Count of Participants; unit: Participants] | 0
Coronary Artery Disease [Count of Participants; unit: Participants] | 10
Hyperlipidemia [Count of Participants; unit: Participants] | 8
Hypertension [Count of Participants; unit: Participants] | 14
Liver Disease [Count of Participants; unit: Participants] | 3
Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 0
Pacemaker/Implantable cardioverter-defibrillator (ICD) [Count of Participants; unit: Participants] | 4
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 3
Prior Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 5
Prior Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] | 5
Prior valve implant [Count of Participants; unit: Participants] | 13
Pulmonary Disease [Count of Participants; unit: Participants] | 2
Pulmonary Hypertension [Count of Participants; unit: Participants] | 12
Stroke [Count of Participants; unit: Participants] | 5
Transient Ischemic Attack (TIA) [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: The primary endpoint for the study will assess the all-cause mortality of the as treated cohort at 30 days compared to a literature derived Performance Goal based on high-risk surgical outcomes for tricuspid repair/replacement. Due to the early termination of the study, the desired statistical power was not attained and thus this comparison analysis was not performed. All-cause mortality is presented below as a number of deaths and percentage of patients only.
Time Frame: At 30 days.
Population: As Treated (AT) Cohort: All subjects who are enrolled and undergo the study procedure (chest incision)
Measure: Count of Participants; unit: Participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 25
Participants | 2

2. Secondary Outcome: Technical Success
Description: Alive, with
  * Successful access, delivery and removal of the delivery systems, and
  * Deployment and correct positioning of the intended device, and
  * No need for additional emergency surgery or re-intervention related to the device or access procedure
Time Frame: Implant Procedure
Population: As Treated (AT) Cohort: all subjects who are enrolled and undergo the study procedure (chest incision)
Measure: Count of Participants; unit: Participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 25
Participants | 22

3. Secondary Outcome: Device Success
Description: Alive, with
  * Original intended device in place, and
  * No additional surgical or interventional procedures related to the device, and
  * Tricuspid Regurgitation (TR) reduction compared to baseline and Tricuspid Valve (TV) gradient ≤ 5 mmHg
Time Frame: At 1 month, 6 months, 1, 2, and 3 years
Population: Implanted Cohort: all subjects who undergo the study procedure (chest incision), receive and retain the investigational device upon leaving the procedure room
  *Count of Participants reflects those subjects who had been implanted, and who had all components of device success
Measure: Count of Participants; unit: Participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 21
Participants
  30 days | 4
  6 months | 3
  1 year | 3
  2 years | 2
  3 years | 0

4. Secondary Outcome: Procedural Success
Description: Device Success, and
  None of the following device or procedure related Serious Adverse Events (SAE):
  * Life threatening bleeding
  * Major vascular or cardiac structural complications requiring intervention
  * Pericardial effusion requiring drainage or surgery (includes tamponade)
  * Stage 2 or 3 acute kidney injury (includes new dialysis).
  * Severe heart failure or hypotension requiring Intravenous (IV) inotrope, ultrafiltration or mechanical circulatory support
  * Prolonged intubation > 48 hours
Time Frame: At 1 month
Population: Implanted Cohort: all subjects who undergo the study procedure (chest incision), receive and retain the investigational device upon leaving the procedure room Denominator reflects those patients who experienced device success and no device or procedure related SAEs
Measure: Count of Participants; unit: Participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 21
Participants | 4

5. Secondary Outcome: Clinical Outcomes [Heart Failure Re-Hospitalization Rates]
Description: Re-hospitalization rates for the underlying condition (heart failure)
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: Kaplan Meier Analysis on Subjects Experiencing Heart Failure Rehospitalization Events
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 25
Percentage of participants
  KM Estimate at 30 days | 100.0 [100.0 to 100.0]
  KM Estimate at 6 months | 91.3 [69.5 to 97.8]
  KM Estimate at 1 year | 85.6 [61.2 to 95.2]
  KM Estimate at 2 years | 72.9 [45.7 to 88.0]
  KM Estimate at 3 years | 72.9 [45.7 to 88.0]

6. Secondary Outcome: Clinical Outcomes [Tricuspid Regurgitation Re-Intervention Rates]
Description: Re-intervention rates for the underlying condition (tricuspid regurgitation)
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: Kaplan Meier Analysis on Subjects Experiencing Re-intervention for Tricuspid Reintervention
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 25
Percentage of participants
  KM Estimate at 30 days | 96.0 [74.8 to 99.4]
  KM Estimate at 6 months | 96.0 [74.8 to 99.4]
  KM Estimate at 1 year | 96.0 [74.8 to 99.4]
  KM Estimate at 2 years | 96.0 [74.8 to 99.4]
  KM Estimate at 3 years | 96.0 [74.8 to 99.4]

7. Secondary Outcome: Clinical Outcomes [Changes in Peripheral Edema]
Description: Change in peripheral edema as assessed by subject weight loss (kilograms) compared to baseline
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: Implanted Cohort: All subjects who underwent the study procedure (chest incision), received and retained the investigational device upon leaving the procedure room
  *Paired Analysis Number of subjects analyzed are those with available paired data at the follow-up
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 22
kg
  Baseline 1 month | 75.1 (14.94)
  1 month | 73.1 (13.34)
  Baseline 6 months: number analyzed (Participants) | 20
  Baseline 6 months | 72.7 (13.25)
  6 months: number analyzed (Participants) | 20
  6 months | 70.2 (11.99)
  Baseline 1 year: number analyzed (Participants) | 17
  Baseline 1 year | 74.3 (13.17)
  1 year: number analyzed (Participants) | 17
  1 year | 71.0 (10.87)
  Baseline 2 years: number analyzed (Participants) | 11
  Baseline 2 years | 76.5 (13.13)
  2 years: number analyzed (Participants) | 11
  2 years | 71.9 (8.80)
  Baseline 3 years: number analyzed (Participants) | 5
  Baseline 3 years | 81.3 (13.93)
  3 years: number analyzed (Participants) | 5
  3 years | 71.8 (11.56)

8. Secondary Outcome: Clinical Outcomes [Change in New York Heart Association (NYHA) Class]
Description: Change in New York Heart Association (NYHA) Class compared to baseline
  Measure Description:
  Measure Description: NYHA Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: Implanted Cohort: All subjects who undergo the study procedure (chest incision), receive and retain the investigational device upon leaving the procedure room
  *Paired Analysis Number of subjects analyzed are those with available paired data at the follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 22
Participants
  Baseline: Class I | 0
  Baseline: Class II | 5
  Baseline: Class III | 12
  Baseline: Class IV | 5
  30 Days: Class I | 2
  30 Days: Class II | 12
  30 Days: Class III | 8
  30 Days: Class IV | 0
  6 months: number analyzed (Participants) | 19
  6 months: Class I | 6
  6 months: Class II | 8
  6 months: Class III | 4
  6 months: Class IV | 1
  1 year: number analyzed (Participants) | 17
  1 year: Class I | 5
  1 year: Class II | 7
  1 year: Class III | 5
  1 year: Class IV | 0
  2 years: number analyzed (Participants) | 11
  2 years: Class I | 5
  2 years: Class II | 5
  2 years: Class III | 0
  2 years: Class IV | 1
  3 years: number analyzed (Participants) | 4
  3 years: Class I | 3
  3 years: Class II | 0
  3 years: Class III | 1
  3 years: Class IV | 0

9. Secondary Outcome: Clinical Outcomes [Change in 6 Minute Walk Test Distance]
Description: Change in 6 minute walk test distance (meters) compared to baseline
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 22
Meters
  Baseline 1 Month: number analyzed (Participants) | 12
  Baseline 1 Month | 328.7 (83.88)
  1 month: number analyzed (Participants) | 12
  1 month | 333.2 (107.90)
  Baseline 6 months: number analyzed (Participants) | 10
  Baseline 6 months | 329.9 (72.49)
  6 months: number analyzed (Participants) | 10
  6 months | 351.6 (77.04)
  Baseline 1 year: number analyzed (Participants) | 8
  Baseline 1 year | 320.9 (76.94)
  1 year: number analyzed (Participants) | 8
  1 year | 353.0 (110.93)
  Baseline 2 years: number analyzed (Participants) | 4
  Baseline 2 years | 322.0 (92.17)
  2 years: number analyzed (Participants) | 4
  2 years | 262.0 (115.85)
  Baseline 3 years: number analyzed (Participants) | 1
  Baseline 3 years | 339.0 (0)
  3 years: number analyzed (Participants) | 1
  3 years | 180.0 (0)

10. Secondary Outcome: Clinical Outcomes [Change in Quality of Life Short Form (SF)-12 Questionnaire]
Description: Change in Quality of Life as assessed by the Short Form (SF)-12 questionnaire compared to baseline The SF-12 is a short survey with 12 questions that results in two scales of mental and physical functioning and overall health related quality of life. The SF-12 Score is scaled from 0-100, with higher scores indicating better physical and mental health functioning.
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 22
score on a scale
  Baseline 1 month | 36.3 (11.14)
  1 month | 39.4 (9.25)
  Baseline 6 months: number analyzed (Participants) | 19
  Baseline 6 months | 37.7 (11.24)
  6 months: number analyzed (Participants) | 19
  6 months | 40.3 (9.75)
  Baseline 1 year: number analyzed (Participants) | 16
  Baseline 1 year | 35.6 (11.03)
  1 year: number analyzed (Participants) | 16
  1 year | 42.7 (12.08)
  Baseline 2 years: number analyzed (Participants) | 10
  Baseline 2 years | 41.0 (10.32)
  2 years: number analyzed (Participants) | 10
  2 years | 44.3 (10.06)
  Baseline 3 years: number analyzed (Participants) | 7
  Baseline 3 years | 40.8 (11.38)
  3 years: number analyzed (Participants) | 7
  3 years | 43.4 (7.41)

11. Secondary Outcome: Clinical Outcomes [Change in Quality of Life Kansas City Cardiomyopathy Questionnaire (KCCQ)]
Description: Change in Quality of Life as assessed by the KCCQ questionnaire compared to baseline The KCCQ is a 12-item questionnaire that quantifies physical limitations, symptoms, self-sufficiency, social interaction and quality of life. The KCCQ scale is 0-100. An increase in the KCCQ-12 score reflects an improvement in symptoms for the subject. A mean difference over time of 5 points on the KCCQ-12 summary score reflects a clinically significant change in heart failure status.
Time Frame: At 1 month, 6 months, 1, 2 and 3 years
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EW Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 22
score on a scale
  Baseline 1 month | 48.7 (31.23)
  1 month | 59.6 (27.68)
  Baseline 6 months: number analyzed (Participants) | 19
  Baseline 6 months | 49.7 (33.11)
  6 months: number analyzed (Participants) | 19
  6 months | 71.9 (28.19)
  Baseline 1 year: number analyzed (Participants) | 16
  Baseline 1 year | 46.2 (34.48)
  1 year: number analyzed (Participants) | 16
  1 year | 70.8 (26.25)
  Baseline 2 years: number analyzed (Participants) | 10
  Baseline 2 years | 60.9 (34.12)
  2 years: number analyzed (Participants) | 10
  2 years | 76.0 (25.48)
  Baseline 3 years: number analyzed (Participants) | 7
  Baseline 3 years | 56.4 (38.97)
  3 years: number analyzed (Participants) | 7
  3 years | 75.9 (22.08)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- EW Tricuspid Transcatheter Repair System: Edwards (EW) Tricuspid Transcatheter Repair System
  EW Tricuspid Transcatheter Repair System: Treatment with the EW Tricuspid Transcatheter Repair System
  As Treated (AT) Cohort: all subjects who are enrolled and undergo the study procedure (chest incision)
Arm/Group | EW Tricuspid Transcatheter Repair System
All-Cause Mortality (participants affected / at risk) | 16/25
Serious Adverse Events (participants affected / at risk) | 20/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EW Tricuspid Transcatheter Repair System (N=25)
Cardiac failure (Cardiac disorders) | 9 (14)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac cirrhosis (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 2 (3)
Septic shock (Infections and infestations) | 2 (2)
Intervertebral discitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 2 (2)
Heart injury (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ventricle rupture (Injury, poisoning and procedural complications) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2)
Anaemia (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (2)
Gastrointestinal haemorrhage (Vascular disorders) | 1 (2)
Intra-abdominal haematoma (Vascular disorders) | 1 (1)
Peripheral artery haematoma (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Rectal haemorrhage (Vascular disorders) | 1 (1)
Syncope (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Nephrogenic anaemia (Renal and urinary disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Intestinal ischemia (Gastrointestinal disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device physical property issue (Product Issues) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EW Tricuspid Transcatheter Repair System (N=25)
Cardiac failure (Cardiac disorders) | 12 (17)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Haematoma muscle (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 2 (2)
Renal failure (Renal and urinary disorders) | 7 (8)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Device related thrombosis (Vascular disorders) | 2 (2)
Epistaxis (Vascular disorders) | 2 (3)
Gastrointestinal haemorrhage (Vascular disorders) | 2 (3)
Shock haemorrhagic (Vascular disorders) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 2 (3)
Septic shock (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 4 (4)
Nerve injury (Nervous system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol: Revision A.G.3 (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02787408/Prot_000.pdf
  • Study Protocol: Revision C (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT02787408/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02787408/SAP_002.pdf